CLINICAL TRIAL: NCT04766385
Title: A Phase 3, Open-label, Single-arm Clinical Study of KHK7791 in Hyperphosphatemia Patients on Peritoneal Dialysis
Brief Title: Clinical Study of KHK7791 in Hyperphosphatemia Patients on Peritoneal Dialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7791-006
Record Dates: First submitted 2021-02-16; First posted 2021-02-23 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Hyperphosphatemia
Keywords: Tenapanor; Hyperphosphatemia; Peritoneal Dialysis
MeSH Terms: conditions — Hyperphosphatemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KHK7791 (Experimental): During the dosing period, subjects administer the study drug (KHK7791 or placebo) twice daily just before meals in a double blind. The starting dose of the study drug is 5 mg at a time, and the dose is adjusted in the range of 5, 10, 20, and 30 mg at a time based on the dose adjustment criteria described in the study protocol. Dosage adjustment is performed step by step.
  Interventions: Drug: KHK7791

INTERVENTIONS:
Drug: KHK7791 — oral administration

SUMMARY:
To evaluate the efficacy of KHK7791 by comparing changes in serum phosphorus levels from baseline values between peritoneal dialysis patients with hyperphosphatemia receiving repeated administration of KHK7791 for 8 weeks and those receiving placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Has voluntarily provided written informed consent to participate in the study.
2. Aged ≥ 20 years (expressed in completed years) at the time of providing informed consent.
3. Stable chronic renal failure patients who have undergone peritoneal dialysis 3 times per week for at least 12 weeks until screening examination.
4. Dialysis conditions, should have been unchanged during the last 2 weeks before screening examination.
5. The prescribed drug and dosage regimen should have been unchanged during the last 2 weeks before screening examination.
6. Serum phosphorus levels should be in the range of ≥ 3.5 and ≤ 7.0 mg/dL at screening examination.
7. If on any vitamin D, calcimimetics regimen, bisphosphonate,calcitonin preparations, selective estrogen receptor modulators or teriparatide preparations then the prescribed drug and dosage regimen should have been unchanged for the last 4 weeks before screening examination.

Exclusion Criteria:

1. Subjects who received concomitant hemodialysis or hemodialysis filtration within 12 weeks before screening examination.
2. Having concurrent or a history of inflammatory bowel disease (IBD) or diarrhea-predominant irritable bowel syndrome
3. History of gastrectomy or enterectomy or having undergone gastrointestinal tract surgery within 3 months before screening examination.
4. Subjects in whom peritonitis, catheter-related infections, catheter dysfunction, etc. are confirmed within 4 weeks before screening examination., and the continuation of peritoneal dialysis is considered to be interfering with the implementation of peritoneal dialysis.
5. Subjects who used anti RANKL preparations within 6 weeks before screening examination.
6. Subjects who used anti-sclerostin antibody preparations within 12 weeks before screening examination.
7. Having concurrent severe heart disease or hepatic impairment.
8. Developed cerebrovascular disease or cardiovascular disease requiring hospitalization within 6 months before screening examination.
9. Subjects who have undergone parathyroid intervention within 24 weeks before screening examination., or subjects who are scheduled to undergo parathyroid intervention between the implementation of the pretest and the completion of the study.
10. Uncontrollable hypertension or diabetes.
11. Scheduled for living donor kidney transplant, change in the mode of dialysis, home hemodialysis, or change in the dialysis center (relocate to another hospital/clinic) during the study period.
12. Any diagnosis of and treatment of malignancy within 5 years before screening examination.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Changes in serum phosphorous levels from baseline values at 8 weeks after the start of administration. | Week 8

SECONDARY OUTCOMES:
Changes in serum phosphorous levels from baseline values at each time point. | Dose period, Week 2, 4, 6, 8, 10, 12, 14, 16.
Achievement/failure of the target serum phosphorus level (serum phosphorus level: ≤ 6.0). | Dose period, Week 2, 4, 6, 8, 10, 12, 14, 16.
Time when the target serum phosphorus level (serum phosphorus level: ≤ 6.0) was achieved. | Dose period, Week 2, 4, 6, 8, 10, 12, 14, 16.
Achievement/failure of the target serum phosphorus level (serum phosphorus level: ≤ 5.5). | Dose period, Week 2, 4, 6, 8, 10, 12, 14, 16.
Time when the target serum phosphorus level (serum phosphorus level: ≤ 5.5) was achieved. | Dose period, Week 2, 4, 6, 8, 10, 12, 14, 16.
Concentrations of such as Ca × P product levels at each time point. | Dose period, Week 2, 4, 6, 8, 10, 12, 14, 16.
Changes of such as Ca × P product levels from baseline values at each time point. | Dose period, Week 2, 4, 6, 8, 10, 12, 14, 16.

CONTACTS AND LOCATIONS:
Locations (1):
- Inoue Hospital, Suita, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nakayama M, Kobayashi S, Kusakabe M, Ohara M, Nakanishi K, Akizawa T, Fukagawa M. Tenapanor for peritoneal dialysis patients with hyperphosphatemia: a phase 3 trial. Clin Exp Nephrol. 2024 Feb;28(2):153-164. doi: 10.1007/s10157-023-02406-1. Epub 2023 Nov 1. PMID 37910313